CLINICAL TRIAL: NCT06094556
Title: A Multicenter, Open Phase I Clinical Study of Safety, Tolerability, Pharmacokinetics, and Efficacy of SHR-1826 for Injection in Patients With Advanced Solid Tumors
Brief Title: An Open Phase I Clinical Trial of SHR-1826 for Injection in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1826-I-101
Record Dates: First submitted 2023-10-16; First posted 2023-10-23 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-1826 (Experimental): Dose escalation; Dose expansion; Therapeutic effect expansion.
  Interventions: Drug: SHR-1826

INTERVENTIONS:
Drug: SHR-1826 — dose is calculated based on the subjects' baseline weight.

SUMMARY:
This is an open, multi-center, dose-escalation/dose-expansion/efficacy expansion phase I clinical study to evaluate the tolerability, safety, PK, and immunogenicity of SHR-1826 in patients with advanced malignant solid tumors, and to preliminatively observe its antitumor efficacy. The whole study was divided into three stages: dose increment, dose extension and therapeutic effect extension.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide a written informed consent.
2. 18-75 years old ，Male or female.
3. ECOG score is 0 or 1.
4. Subjects with advanced or metastatic solid tumors that have been documented by histopathology and are not responding to or tolerated by standard treatment, or have no effective standard treatment options.
5. Have at least one measurable lesion according to RECIST v1.1 criteria.
6. Expected survival ≥3 months .
7. With good vital organ function.
8. Contraception.

Exclusion Criteria:

1. With untreated or active Central nervous system (CNS) tumor metastasis. Subjects with a history or current history of meningeal metastasis.
2. Previous or co-existing malignant tumors.
3. Spinal cord compression that was not treated radically by surgery and/or radiotherapy was excluded.
4. Patients with uncontrolled tumor-related pain.
5. Received systemic antitumor therapy 4 weeks before starting study treatment; Previously receiving small molecule targeted therapy, the interval of not less than 5 half-lives of the drug can be enrolled.
6. Previously received antibody-coupled drug therapy.
7. Have undergone major surgery other than diagnosis or biopsy within 28 days prior to initial dosing; Minor traumatic surgery within 7 days prior to first dosing.
8. First study subjects receiving >30Gy non-radical chest radiation within 28 days prior to administration, >30Gy chest radiation within 24 weeks prior to first administration, and ≤30Gy palliative radiation within 14 days prior to first administration;If previously received radioisotope therapy, the interval of not less than 5 half-lives of the isotope drug can be included.
9. Is participating in another clinical study or the time of first administration is less than 4 weeks from the end of the previous clinical study (last administration), or the 5 half-life of the investigational drug, whichever is the older.
10. The AE caused by previous anti-tumor therapy did not recover to CTCAE v5.0 grade evaluation ≤1.
11. Other severe lung diseases that may interfere with the detection or management of drug-related pulmonary toxicity within the first three months of administration that significantly affect respiratory function; Any autoimmune, connective tissue, or inflammatory disease with lung involvement; Prior left or right total lung resection.
12. Pleural effusion, ascites, or pericardial effusion requiring intervention occurred within 2 weeks prior to the first dose.
13. Have an active autoimmune disease, or other acquired (HIV infection), congenital immunodeficiency disease, or a history of organ transplantation.
14. Have poorly controlled or severe cardiovascular disease.
15. Known hereditary or acquired bleeding and thrombotic tendencies, and clinically significant bleeding symptoms and arterial/venous thrombosis events in the 3 months prior to the first dose.
16. Untreated active hepatitis.
17. Subjects who had a severe infection within 30 days prior to the first dose; Patients with active pulmonary tuberculosis infection within 1 year prior to enrollment were found by medical history or CT examination, or had a history of active pulmonary tuberculosis infection more than 1 year ago but had not received regular treatment.
18. Live attenuated vaccine should be administered within 30 days prior to the first dose.
19. Female subjects who are pregnant, breastfeeding, or planning to become pregnant during the study period.
20. Known allergy to any component or excipient of the SHR-1826 product.
21. The presence of other serious physical or mental illnesses or abnormalities in laboratory tests that may increase the risk of participation in the study, or interfere with the study results, as well as conditions that the investigator deems inappropriate to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-12-25 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity | 21 Days
  evaluate the safety in the doses escalation
Maximum tolerated dose or Maximum-administered dose | Approximately 1 year
  evaluate the safety in the doses escalation
Recommended Phase 2 dose (RP2D) | Approximately 2 years
  evaluate the safety and curative effect in the doses escalation

SECONDARY OUTCOMES:
Maximum concentration (Cmax) of SHR-1826 | Approximately 2 years
  To evaluate the pharmacokinetic characteristics of SHR-1826
Time to maximum concentration (Tmax) of SHR-1826 | Approximately 2 years
  To evaluate the pharmacokinetic characteristics of SHR-1826
Areas under the concentration-time curve from time zero to the time of last quantifiable concentration (AUClast) of SHR-1826 | Approximately 2 years
  To evaluate the pharmacokinetic characteristics of SHR-1826
Areas under the concentration-time curve from time zero extrapolated to infinity (AUCinf) of SHR-1826 | Approximately 2 years
  To evaluate the pharmacokinetic characteristics of SHR-1826
Half-life (t1/2) of SHR-1826 | Approximately 2 years
  To evaluate the pharmacokinetic characteristics of SHR-1826
Mean retention times (MRT) of SHR-1826 | Approximately 2 years
  To evaluate the pharmacokinetic characteristics of SHR-1826
Clearance rate (CL) of SHR-1826 | Approximately 2 years
  To evaluate the pharmacokinetic characteristics of SHR-1826
Volume of distribution at the steady state (Vss) of SHR-1826 | Approximately 2 years
  To evaluate the pharmacokinetic characteristics of SHR-1826
Anti-drug antibody of SHR-1826 | Approximately 2 years
  To evaluate the pharmacokinetic characteristics of SHR-1826
Objective response rate (ORR) | Approximately 2 years
  Preliminary evaluation of the effectiveness of SHR-1826
Duration of response (DoR) | Approximately 2 years
  Preliminary evaluation of the effectiveness of SHR-1826
Disease control rate (DCR) | Approximately 2 years
  Preliminary evaluation of the effectiveness of SHR-1826
Progression free survival (PFS) | Approximately 2 years
  Preliminary evaluation of the effectiveness of SHR-1826
Overall survival (OS) | Approximately 2 years
  Preliminary evaluation of the effectiveness of SHR-1826

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided